CLINICAL TRIAL: NCT05507463
Title: A Phase I, Double-blind, Placebo-controlled, Single and Multiple Intravenous Dose, Safety, Tolerability and Pharmacokinetic Study of KBP-7072 in Healthy Male and Female Subjects
Brief Title: Study of KBP-7072 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBP7072-1-004
Record Dates: First submitted 2022-06-24; First posted 2022-08-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — kbp-7072

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KBP-7072 (Experimental): Proposed dose levels for Part A: 25, 50, 100, 150 and 200mg KBP-7072. Proposed dose levels for Part B: 50 and 100mg. Administration route is intravenous infusion.
  Interventions: Drug: KBP-7072
- Placebo (Placebo Comparator): Placebo for intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KBP-7072 — KBP-7072
  Arms: KBP-7072
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, single and multiple IV dose study conducted in two parts. Part A (SAD) will comprise an ascending single dose, sequential group design. Each subject will participate in 1 treatment period only. Subjects will reside at the study site from check-in on Day -1 (the day before dosing) to discharge on Day 8. In Part A, serial blood and urine collections will be obtained on Day 1 pre-dose through 168 hours post start of infusion for analysis of plasma and urine concentrations of KBP-7072 and KBP-6079. Safety will be monitored through recording of adverse events, clinical laboratory evaluations, vital sign measurements, 12-lead ECG and physical examination findings. Part B (MAD) will comprise an ascending multiple dose, sequential group study. Each subject will participate on one treatment period only and reside at the study site from check-in on Day -1 until discharge on Day 17. In Part B, serial blood and urine collections will be obtained on Day 1 pre-dose through 24 hours post start of infusion and on Day 10 pre-dose through 168 hours post start of infusion for analysis of plasma and urine concentrations of KBP-7072 and KBP-6079. Trough blood sample collections for analysis of plasma concentrations of KBP-7072 and KBP-6079 will be obtained pre-dose on Days 3, 4, 5, 6, 7, 8 and 9. Safety will be monitored through recording of adverse events, clinical laboratory evaluations, vital sign measurements, 12-lead ECG and physical examination findings.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30 kg/m2 at the time of screening
* In good health, determined b no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements and clinical laboratory evaluations
* Females of nonchildbearing potential defined as permanently sterile or postmenopausal.

Males will agree to use contraception.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine or psychiatric disorder as determined by the investigator.
* Abnormal results of ophthalmologic examination within 3 months prior to dosing self-reported by subject.
* Supine systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg.
* Triglycerides > 200 mg/dL
* Total cholesterol > 240 mg/dL or LDL >190 mg/dL or HDL < 40 mg/dL
* Positive urine drug screen at screening or check-in or positive blood alcohol test result at check-in.
* Positive hepatitis panel and/or positive HIV test
* Administration of a Covid-19 vaccine in the past 28 days prior to dosing
* Interpretation of liver ultrasound with presence of fatty liver disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, with abnormal laboratory test results, abnormal ECGs, abnormal vital signs, and abnormal physical examinations | Time Frame: SAD 1- 7 days and MAD 1-17 days
  Safety Assessment evaluated through adverse events, laboratory evaluations, vital signs, ECGs, and physical examination.

SECONDARY OUTCOMES:
Pharmacokinetics Parameters :AUC from time 0 extrapolated to infinity (AUC0-∞) | SAD Day 1 predose (within the 30 minutes prior to dosing) and at 5, 15,30,45 minutes and at 1,1.5,2,4,6,10,12,24 (day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7) and 168 (Day 8) hour(s) post start of infusion
  AUC from time 0 extrapolated to infinity (AUC0-∞)
Pharmacokinetics Parameters: Area under the plasma concentration-time curve (AUC) from time zero to time of last quantifiable concentration (AUC0-tlast), | SAD Day 1 predose (within the 30 minutes prior to dosing) and at 5, 15,30,45 minutes and at 1,1.5,2,4,6,10,12,24 (day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7) and 168 (Day 8) hour(s) post start of infusion
  Area under the plasma concentration-time curve (AUC) from time zero to time of last quantifiable concentration (AUC0-tlast) - Plasma
Pharmacokinetics Parameters: AUC over a dosing interval (AUC0-τ), from time zero to time of last quantifiable concentration (AUC0-tlast)from time zero to time of last quantifiable concentration (AUC0-tlast) | MAD samples will be collected on Day 1 pre-dose and at 5, 15, 30, 45 minutes, and at 1, 1.5, 2, 4, 6, 10, 12, 24 (Day 2) hours, pre-dose samples at 48 (Day 3), 72 (Day 4), 96 (Da
  AUC over a dosing interval (AUC0-τ) - Plasma
Pharmacokinetics Parameters: Maximum observed plasma concentration (Cmax) | SAD Day 1 predose (within the 30 minutes prior to dosing) and at 5, 15,30,45 minutes and at 1,1.5,2,4,6,10,12,24 (day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7) and 168 (Day 8) hour(s) post start of infusion
  Maximum observed plasma concentration (Cmax) - Plasma
Pharmacokinetics Parameters: time of the maximum observed plasma concentration (Tmax) | SAD Day 1 predose (within the 30 minutes prior to dosing) and at 5, 15,30,45 minutes and at 1,1.5,2,4,6,10,12,24 (day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7) and 168 (Day 8) hour(s) post start of infusion
  Time of the maximum observed plasma concentration (Tmax) - Plasma
Pharmacokinetics Parameters: apparent terminal elimination half-life (t1/2) | SAD Day 1 predose (within the 30 minutes prior to dosing) and at 5, 15,30,45 minutes and at 1,1.5,2,4,6,10,12,24 (day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7) and 168(Day 8) hour(s) post start of infusion
  Apparent terminal elimination half-life (t1/2) - Plasma
Pharmacokinetics Parameters: observed accumulation ratio based on AUC0-τ (ARAUC0-τ) | MAD samples will be collected on Day 1 pre-dose and at 5, 15, 30, 45 minutes, and at 1, 1.5, 2, 4, 6, 10, 12, 24 (Day 2) hours, pre-dose samples at 48 (Day 3), 72 (Day 4), 96 (Da
  Observed accumulation ratio based on AUC0-τ (ARAUC0-τ) - Plasma
Pharmacokinetics Parameters: amount of drug excreted in urine (Ae) | SAD Day 1 predose (within the 30 minutes prior to dosing) and at 5, 15,30,45 minutes and at 1,1.5,2,4,6,10,12,24 (day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7) and 168(Day 8) hour(s) post start of infusion
  Amount of drug excreted in urine (Ae) - Urine

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, Principal Investigator — Parexel
Locations (1):
- Parexel International - Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No